CLINICAL TRIAL: NCT00659282
Title: Observational Study of Safety and Effectiveness of NovoMix® 30 (Biphasic Insulin Aspart) for the Treatment of Diabetes Mellitus
Brief Title: Observational Study of Safety and Effectiveness of NovoMix® 30 for the Treatment of Diabetes
Acronym: IMPROVE™
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1766
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: biphasic insulin aspart
  Interventions: Drug: biphasic insulin aspart

INTERVENTIONS:
Drug: biphasic insulin aspart — Start dose and frequency to be prescribed by the physician as a result of a normal clinical evaluation.
  Other Names: BIASP; NovoMix 30; NovoLog Mix 70/30

SUMMARY:
This study is conducted in Asia, Europe, Japan and North America. The aim of this observational study is to evaluate the safety and effectiveness while using NovoMix® 30 during 26 weeks under normal clinical practice, in the countries participating in the study. The primary outcome is the incidence of major hypoglycaemic events reported as serious adverse drugs reaction conditions on hypoglycaemic events.

ELIGIBILITY:
Inclusion Criteria:

* Age according to approved label and physician discretion
* Type 2 diabetes including newly-diagnosed subjects who have never received insulin or an insulin analogue before

Exclusion Criteria:

* Subjects who previously enrolled in this study
* Subjects who are unlikely to comply with protocol requirements
* Hypersensitivity to biphasic insulin aspart or to any of the excipients
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within next 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from both general and speciality practice settings who have been deemed appropriate to receive NovoMix® 30 as new treatment and as part of routine out-patient care by the prescribing physician.
Sampling Method: Non-Probability Sample
Enrollment: 57610 (Actual)
Dates: Start 2006-09-11 (Actual); Primary Completion 2008-11-15 (Actual); Study Completion 2008-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence of major hypoglycaemic events reported as serious adverse drug reactions | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (11):
- Novo Nordisk Investigational Site, Mississauga, Canada
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China
- Novo Nordisk Investigational Site, Vouliagment, Greece
- Novo Nordisk Investigational Site, Bangalore, India
- Novo Nordisk Investigational Site, Tehran, Iran
- Novo Nordisk Investigational Site, Rome, Italy
- Novo Nordisk Investigational Site, Tokyo, Japan
- Novo Nordisk Investigational Site, Warsaw, Poland
- Novo Nordisk Investigational Site, Moscow, Russia
- Novo Nordisk Investigational Site, Riyadh, Saudi Arabia
- Novo Nordisk Investigational Site, Seoul, South Korea

REFERENCES:
- [Result] Valensi P, Benroubi M, Borzi V, Gumprecht J, Kawamori R, Shaban J, Shah S, Shestakova M, Wenying Y; IMPROVE Study Group Expert Panel. The IMPROVE study--a multinational, observational study in type 2 diabetes: baseline characteristics from eight national cohorts. Int J Clin Pract. 2008 Nov;62(11):1809-19. doi: 10.1111/j.1742-1241.2008.01917.x. Epub 2008 Sep 22. PMID 18811598
- [Result] Valensi P, Benroubi M, Borzi V, Gumprecht J, Kawamori R, Shaban J, Shah S, Shestakova M, Wenying Y; IMPROVE Study Group Expert Panel. Initiating insulin therapy with, or switching existing insulin therapy to, biphasic insulin aspart 30/70 (NovoMix 30) in routine care: safety and effectiveness in patients with type 2 diabetes in the IMPROVE observational study. Int J Clin Pract. 2009 Mar;63(3):522-31. doi: 10.1111/j.1742-1241.2009.02002.x. Epub 2009 Jan 27. PMID 19187170
- [Result] Wenying Y, Benroubi M, Borzi V, Gumprecht J, Kawamori R, Shaban J, Shah S, Shestakova M, Ligthelm R, Valensi P; IMPROVE Study Group Expert Panel. Improved glycaemic control with BIAsp 30 in insulin-naive type 2 diabetes patients inadequately controlled on oral antidiabetics: subgroup analysis from the IMPROVE study. Curr Med Res Opin. 2009 Nov;25(11):2643-54. doi: 10.1185/03007990903276745. PMID 19751116
- [Result] Yang W, Gao Y, Liu G, Chen L, Fu Z, Zou D, Feng P, Zhao Z. Biphasic insulin aspart 30 as insulin initiation or replacement therapy: the China cohort of the IMPROVE study. Curr Med Res Opin. 2010 Jan;26(1):101-7. doi: 10.1185/03007990903364640. PMID 19916705
- [Result] Gumprecht J, Benroubi M, Borzi V, Kawamori R, Shaban J, Shah S, Shestakova M, Wenying Y, Ligthelm R, Valensi P; IMPROVE Study Group Expert Panel. Intensification to biphasic insulin aspart 30/70 (BIAsp 30, NovoMix 30) can improve glycaemic control in patients treated with basal insulins: a subgroup analysis of the IMPROVE observational study. Int J Clin Pract. 2009 Jun;63(6):966-72. doi: 10.1111/j.1742-1241.2009.02064.x. PMID 19504715
- [Result] Ishii H, Iwase M, Seino H, Shuto Y, Atsumi Y. Assessment of quality of life in patients with type 2 diabetes mellitus before and after starting biphasic insulin aspart 30 (BIAsp 30) therapy: IMPROVE study in Japan. Curr Med Res Opin. 2011 Mar;27(3):643-50. doi: 10.1185/03007995.2010.551760. Epub 2011 Jan 21. PMID 21250861
- [Result] Shah S, Benroubi M, Borzi V, Gumprecht J, Kawamori R, Shaban J, Shestakova M, Wenying Y, Valensi P; IMPROVE Study Group Expert Panel. Safety and effectiveness of biphasic insulin aspart 30/70 (NovoMix 30) when switching from human premix insulin in patients with type 2 diabetes: subgroup analysis from the 6-month IMPROVE observational study. Int J Clin Pract. 2009 Apr;63(4):574-82. doi: 10.1111/j.1742-1241.2009.02012.x. Epub 2009 Feb 5. PMID 19210701
- [Result] Valensi P, Shaban J, Benroubi M, Kawamori R, Borzi V, Shah S, Wenying Y, Prusty V, Hansen JB, Gumprecht J; IMPROVE Study Expert Panel. Predictors of achieving HbA(1c) <7% and no hypoglycaemia 6 months after initiation of biphasic insulin aspart 30 in patients with type 2 diabetes in the IMPROVE study. Curr Med Res Opin. 2013 Jun;29(6):601-9. doi: 10.1185/03007995.2013.786692. Epub 2013 Apr 12. PMID 23488447
- [Result] Valensi P, Husemoen LLN, Weatherall J, Monnier L. Association of postprandial and fasting plasma glucose with HbA1c across the spectrum of glycaemic impairment in type 2 diabetes. Int J Clin Pract. 2017 Dec;71(12):e13041. doi: 10.1111/ijcp.13041. No abstract available. PMID 29283504
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com